CLINICAL TRIAL: NCT06420154
Title: An Exploratory Clinical Study to Evaluating the Safety and Efficacy of Infusiing Anti-CD19-CAR-T Cells Injection (Anti-CD19-CAR-T Cells) in Patients With Relapsed/Refractory Autoimmune Diseases
Brief Title: The Safety and Efficacy of Anti-CD19 CAR-T Cells in Patients With Relapsed/Refractory Autoimmune Diseases
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Shanghai First Song Therapeutics Co., Ltd (Industry)
Responsible Party: Principal Investigator, Li Sun, Professor and Chief Physician, Head of the Department of Rheumatology and Immunology, The First Affiliated Hospital of Wenzhou Medical University, First Affiliated Hospital of Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19-CN-A4
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Systemic Lupus Erythematosus (SLE); Sjogren's Syndrome; Systemic Sclerosis; Inflammatory Myopathy; ANCA Associated Vasculitis; Antiphospholipid Syndrome
Keywords: CAR T; CD19; Autoimmune Diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Sjogren's Syndrome; Scleroderma, Systemic; Myositis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Antiphospholipid Syndrome; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Biological: anti-CD19-CAR-T cells

INTERVENTIONS:
Biological: anti-CD19-CAR-T cells — The subjects received infusions of anti-CD19 CAR-T cells following completion of lymphodepleting preconditioning chemotherapy.
  Dosage：1×10^5 cells/Kg; 3×10^5 cells/Kg; 1×10^6 cells/Kg
  frequency：single infusion

SUMMARY:
This is an investigator-initiated trial to evaluate the safety and efficacy of anti- CD19-CAR-T cells in the relapse or refractory autoimmune diseases.

DETAILED DESCRIPTION:
This is an investigator-initiated trial to evaluate the safety and efficacy of anti- CD19-CAR-T cells in the relapse or refractory autoimmune diseases.

Study intervention consists of a single infusion of CAR-transduced autologous T cells administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide.

Interim analysis will be performed when the last participant finishes the visit of 12 weeks after CAR-T cells infusion.

ELIGIBILITY:
Common Inclusion Criteria:

1. Voluntarily participate in clinical research. The person or legal guardian fully understands and informs the research and signs the informed consent form (ICF), and is willing to follow and complete all trial procedures;
2. Aged 18-65 years old;
3. ECOG score ≤ 2 points;
4. Expected survival period is at least 12 weeks;
5. Have good intravenous access (for apheresis) and have no other contraindications to blood cell separation;
6. When screening patients, laboratory tests must meet the following requirements and they must not have received cell growth factors within 7 days before screening hematology assessment (long-acting colony-stimulating factor (G-CSF/PEG-CSF) requires an interval of 2 weeks):

<!-- -->

1. Absolute neutrophil count ≥1.0×10^9/L;
2. Hemoglobin ≥60 g/L (without red blood cell transfusion within 14 days);
3. Platelets ≥50×10^9/L;
4. Absolute lymphocytes (ALC) ≥ 0.5×10^9/L;
5. Serum total bilirubin ≤1.5×upper limit of normal (ULN);
6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN;
7. Creatinine <1.5×ULN and endogenous creatinine clearance ≥60 mL/min. 7. The cardiac ejection fraction is ≥45%, echocardiography (ECHO) confirms that there is no pericardial effusion (except for a small amount or physiological), and the electrocardiogram results have no clinical significance; 8. Baseline oxygen saturation >92% under non-oxygenation conditions; 9. Women of childbearing age must have a negative serum or urine pregnancy test report (women who have undergone surgical sterilization or women who are at least 2 years postmenopausal are not considered women of childbearing potential).

Common Exclusion Criteria:

1. Have active central nervous system diseases, such as epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving the central nervous system;
2. Fungal, bacterial, viral or other infections exist or are suspected and are not controlled or require intravenous antibiotic treatment; simple urinary tract infections and uncomplicated bacterial pharyngitis are allowed;
3. Suffering from hepatitis B (hepatitis B virus surface antigen and hepatitis B DNA >1000 copies/ml) or hepatitis C (positive hepatitis C antibody test); syphilis infection (antibody positive); human immunodeficiency virus (HIV) infection;
4. Past medication:

<!-- -->

1. CD19 targeted therapy;
2. Inject live vaccines within 4 weeks before enrollment;
3. Immunosuppressive antibodies (such as anti-CD20, anti-tumor necrosis factor, anti-interleukin 6 or anti-interleukin 6 receptor) used within 4 weeks before enrollment;
4. Use immunostimulatory or immune enhancer treatment (such as tacrolimus, cyclosporine, interferon-α, interferon-β, IL-2) within the 5 half-lives before apheresis;
5. Have used systemic cytotoxic drugs within 2 weeks before enrollment, including daily or weekly low-dose maintenance chemotherapy (cyclophosphamide, ifosfamide, bendamustine, clotrexate or Melphalan, vincristine, etc.);
6. Long-acting growth factors within 14 days before apheresis (such as pegfilgrastim) or short-acting growth factors within 5 days before apheresis or drugs used for cell mobilization (such as granulocyte colony-stimulating factor/non- Gestin, Plexafor);
7. The use of pharmacological doses of corticosteroids (>10 mg/day of prednisone or equivalent doses of other corticosteroids) and other immunosuppressive drugs must be avoided within 4 days before enrollment.

5. Have a history of myocardial infarction, cardiac angioplasty or stent implantation, unstable angina or other clinically significant heart diseases within 12 months before enrollment; 6. History of genetic syndromes associated with bone marrow failure, such as Fanconi anemia, Kosterman syndrome, Swachmann-Diamond syndrome, etc.; 7. History of symptomatic deep vein thrombosis or pulmonary embolism requiring systemic anticoagulation within 6 months before enrollment. Subjects need to take prophylactic anticoagulant drugs; 8. Have suffered from other malignant tumors in the past or at the same time (except for basal cell carcinoma of the skin, carcinoma in situ of the breast/cervix and other malignant tumors that have been effectively controlled without treatment in the past five years); 9. Use of other investigational pharmaceutical products within 30 days before screening; 10.Women of childbearing age who are pregnant or breastfeeding (because chemotherapy has potentially dangerous effects on the fetus or baby); 11.Male and female subjects who are unwilling to undergo birth control within 6 months from the signing of the informed consent form to the completion of the last administration of the study drug; 12.Any medical activity that may interfere with the evaluation of the safety or efficacy of the study; 13.According to the investigator's judgment, the subject is unlikely to complete all study visits or procedures required by the protocol, including follow-up visits or comply with the requirements for participation in the study; 14.Those who have used any CAR-T cell products or other genetically modified T cell therapies in the past.

Specific inclusion/exclusion criteria:

Relapsed and refractory systemic lupus erythematosus： Inclusion criteria：

1. Comply with the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) SLE classification criteria;
2. In the moderate to severe active stage of the disease, SELENA-SLEDAI score >6;
3. And have at least one British Island Lupus Assessment Group Index (BILAG-2004) Category A (severe performance) or two Category B (moderate performance) organ scores, or both;
4. Definition of relapse and refractory: Conventional treatment is ineffective or disease activity reappears after remission. The definition of routine treatment: the use of glucocorticoids (more than 1 mg/Kg/d) and cyclophosphamide, and any one or more of the following immunomodulatory drugs for more than 6 months: antimalarial drugs, azathioprine, mycophenolate mofetil , methotrexate, leflunomide,tacrolimus,cyclosporine, and biological agents including rituximab, belimumab, tatacept, etc.

Exclusion criteria:

1. Combined with neuropsychiatric lupus;
2. Thrombotic thrombocytopenic purpura (TTP)/microthrombotic vasculopathy (TMA).

Relapsed and Refractory Sjogren's Syndrome Inclusion criteria：

1. Meet the 2002 AECG criteria or the 2016 ACR/EULAR classification criteria for primary sjogren's syndrome;
2. Definition of relapse and refractory: Conventional treatment is ineffective or disease activity reappears after remission. The definition of routine treatment: the use of glucocorticoids (more than 1 mg/Kg/d) and cyclophosphamide, and any one or more of the following immunomodulatory drugs for more than 6 months: antimalarial drugs, azathioprine, mycophenolate mofetil , methotrexate, leflunomide, tacrolimus, cyclosporine, and biological agents including rituximab, belimumab, tatacept, etc.

Exclusion criteria:

1. Combined with liver cirrhosis;
2. Combined with aplastic anemia (AA), myelodysplastic syndrome (MDS) or other myeloproliferative diseases (MPD);
3. Drug-induced thrombocytopenia;
4. Thrombotic thrombocytopenic purpura (TTP)/microthrombotic vasculopathy (TMA).

Relapsed, Refractory/Progressive Diffuse Scleroderma

Inclusion criteria： 1.Comply with the 2013 ACR classification criteria for scleroderma and comply with diffuse manifestations; 2.Combined with interstitial pneumonia: chest HRCT shows interstitial changes with ground glass exudation and the predicted value of FVC or DLCO in pulmonary function testing is <70%; 3.Definition of relapse and refractory: Conventional treatment is ineffective or disease activity reappears after remission. The definition of routine treatment: the use of glucocorticoids (more than 1 mg/Kg/d) and cyclophosphamide, and any one or more of the following immunomodulatory drugs for more than 6 months: antimalarial drugs, azathioprine, mycophenolate mofetil , methotrexate, leflunomide, tacrolimus, cyclosporine and biological agents including rituximab, belimumab, tatacept, etc.; 4.Definition of progress:

1. Definition of skin progression: mRSS increase >10%;
2. Definition of lung disease progression: FVC decreases by 10%, or FVC decreases by 5% and DLCO decreases by 15% (OMERACT progression).

   Exclusion criteria:
   1. New York heart function class IV;
   2. There is moderate to severe pulmonary hypertension (mean pulmonary artery pressure on echocardiography >40 mmHg);
   3. FVC <45% predicted value;
   4. DLCO <40% predicted value;
   5. Significant abnormalities on HRCT are not caused by SSc;
   6. Persistent unexplained hematuria (5 red blood cells under high power) or creatinine clearance <40ml/min;
   7. Patients who have had autologous stem cell transplantation in the past;
   8. There are signs of renal crisis;
   9. Active antral vasodilation.

   Relapsed Refractory/Progressive Inflammatory Myopathy

   Inclusion criteria： 1.Comply with the 2017 EULAR/ACR classification criteria for inflammatory myopathies (including DM, PM, ASS and NM); 2.For those with muscle involvement, the MMT-8 score is lower than 142 and there are at least two abnormal findings in the following five core measurements (PhGA, PtGA or extramuscular disease activity score ≥ 2 points; HAQ total score ≥ 0.25; muscle enzymes level is 1.5 times the upper limit of the normal range); 3.Myositis antibody positive; 4.Definition of relapse and refractory: Conventional treatment is ineffective or disease activity reappears after remission. The definition of routine treatment: the use of glucocorticoids (more than 1 mg/Kg/d) and cyclophosphamide, and any one or more of the following immunomodulatory drugs for more than 6 months: antimalarial drugs, azathioprine, mycophenolate mofetil , methotrexate, leflunomide, tacrolimus, cyclosporine, and biological agents including rituximab, belimumab, tatacept, etc.

   5.Definition of progressive: Rapidly progressive interstitial pneumonia occurring in a short period of time.

   Exclusion criteria:
   1. Drug-induced myositis
   2. Inclusion body myositis;
   3. Tumor-related myositis (myositis occurring within 2 years after tumor diagnosis).

   Relapsed and Refractory ANCA-Associated Vasculitis

   Inclusion criteria：

   1.Meet the 2022 ACR/EULAR diagnostic criteria for ANCA vasculitis, including microscopic polyangiitis, granulomatosis with polyangiitis, and eosinophilic granulomatosis with polyangiitis; 2.Positive ANCA-related antibodies (MPO-ANCA or PR3-ANCA positive); 3.Birmingham Vasculitis Activity Score (BVAS) ≥15 points (total score 63 points), indicating active vasculitis; 4.There must be at least one major item, at least 3 minor items, or at least two renal items in the BVAS assessment: hematuria and proteinuria; 5.Definition of relapse and refractory: Conventional treatment is ineffective or disease activity reappears after remission. The definition of routine treatment: the use of glucocorticoids (more than 1 mg/Kg/d) and cyclophosphamide, and any one or more of the following immunomodulatory drugs for more than 6 months: antimalarial drugs, azathioprine, mycophenolate mofetil , methotrexate, leflunomide, tacrolimus, cyclosporine and biological agents including rituximab, belimumab, tatacept, etc.;

   Exclusion criteria:

   1.Estimated glomerular filtration rate (eGFR) <15 mL/min/1.73 m2; 2.If the patient has alveolar hemorrhage, invasive pulmonary ventilation is required and the duration is expected to exceed the screening time; 3.Dialysis or plasma exchange is required during the screening period; 4.Have received a kidney transplant.

   Relapsed/Refractory/Catastrophic Antiphospholipid Syndrome

   Inclusion criteria：
   1. Meet the diagnostic criteria for primary antiphospholipid syndrome revised in Sydney in 2006;
   2. Positive medium-to-high titer phospholipid antibodies (LA, B2GP1 or acL IgG/IgM, more than two positive tests within 12 weeks);
   3. Definition of relapse and refractory: use of warfarin anticoagulation or standard treatment instead of vitamin K antagonists (i.e., maintenance of the INR required for treatment) or use of standard therapeutic doses of low molecular weight heparin (LMWH), as well as use of hormones and cyclophosphamide treatment Recurrence of thrombosis;
   4. Catastrophic antiphospholipid syndrome requires the following four criteria:

   <!-- -->

   1. Involving three or more organs, systems and/or tissues;
   2. Symptoms appear within 1 week;
   3. Histology confirms small blood vessel obstruction in at least one organ or tissue;
   4. aPL positive.

   Exclusion criteria:
   1. Obstetric APS;
   2. APS merged with other CTDs;
   3. APS involves the nervous system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-05-27 (Estimated); Primary Completion 2027-05-27 (Estimated); Study Completion 2027-05-27 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity | Up to 28 days from CAR-T infusion
  Percentage of patients receiving CAR-T cells who experience dose-limiting toxicities (DLTs).
Laboratory abnormalities and type, frequency and severity of adverse events | Up to1 year from CAR-T infusion
  Safety assessments are conducted using the NCI-CTCAE version 5.0 standards (CRS and neurotoxicity will be graded according to ASTCT/ ASBMT grading criteria)
Proportion of patients for whom a CAR-T cell product could be prepared | Up to 4 days from apheresis
  Percentage of subjects for whom the desired dose of anti-CD19 -CAR-T cells can be successfully manufactured

CONTACTS AND LOCATIONS:
Overall Officials: LI Sun, Master's, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Due to concerns regarding the security of patient personal information.